CLINICAL TRIAL: NCT05211154
Title: A Randomized, Parallel-Group, Single-Attack, Open-Label Study to Evaluate the Efficacy of Diclofenac Potassium and Rimegepant for the Acute Treatment of Migraine (ATOM)
Brief Title: Evaluation of the Efficacy of Diclofenac Potassium and Rimegepant for the Acute Treatment of Migraine
Acronym: ATOM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Issues with recruitment
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Messoud Ashina, MD, Professor, Danish Headache Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 260221; 2021-001057-31 (EudraCT Number)
Record Dates: First submitted 2022-01-11; First posted 2022-01-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Migraine With Aura; Migraine Without Aura
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura | interventions — Diclofenac; rimegepant sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diclofenac Potassium (soluble) (Experimental): 50 mg diclofenac potassium taken orally once
  Interventions: Drug: Diclofenac Potassium 50Mg/Pkt Oral Pwdr
- Rimegepant (Active Comparator): 75 mg rimegepant taken orally once
  Interventions: Drug: Rimegepant 75 MG

INTERVENTIONS:
Drug: Diclofenac Potassium 50Mg/Pkt Oral Pwdr — Treatment for an acute, moderate to severe migraine attack
  Other Names: Voltfast
  Arms: Diclofenac Potassium (soluble)
Drug: Rimegepant 75 MG — Treatment for an acute, moderate to severe migraine attack
  Arms: Rimegepant

SUMMARY:
In a real-world population of adults with migraine, the investigators would like to investigate whether 50 mg diclofenac potassium is non-inferior to 75 mg rimegepant in terms of pain freedom at 2 hours after drug intake.

DETAILED DESCRIPTION:
The study design is a randomized, open-label, parallel-group, single-attack study with 50 mg diclofenac potassium and 75 mg rimegepant. 645 patients with migraine with or without aura according to the third edition of the International Classification of Headache Disorders (ICHD-3) will be included.

Each subject will randomly be allocated to one treatment, and given 42 days to treat a single qualifying migraine attack of moderate to severe intensity.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures.
* Aged 18 to 65 years upon entry into screening
* History of migraine (with or without aura) for greater than or equal to 12 months before screening according to the ICHD-3 criteria based on medical records and/or patient self-report.
* Not more than 12 attacks per month with moderate to severe headache pain in each of the previous 3 months.

Exclusion Criteria:

Disease Related

* Greater than 50 years of age at migraine onset
* History of cluster headache or hemiplegic migraine headache
* Inability to differentiate between migraine from other headaches
* Has taken medication for acute treatment of headache (including acetaminophen, nonsteroidal anti-inflammatory drugs (NSAIDs), triptans, ergotamine, opioids, or combination analgesics) on 10 or more days per months in the previous 3 months
* Has a history of migraine aura with diplopia or impairment of levels of consciousness, hemiplegic migraine, or retinal migraine.
* Required hospital treatment of a migraine attack 3 or more times in the previous 6 months.

Other Medical Conditions

* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* Has a chronic non-headache pain condition requiring daily pain medication
* Has a history of any prior gastrointestinal conditions (e.g., diarrhea syndromes, inflammatory bowel disease) that may affect the absorption or metabolism of investigational product; participants with prior gastric bariatric interventions which have been reversed are not excluded.
* Has a history of malignancy in the prior 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer.
* History or evidence of any other clinically significant disorder, condition or disease (except for those outlined above) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion

Medication related

* Start of new preventive migraine treatment within the last two months
* Change in dosage of ongoing preventive migraine treatment within the last two months
* Current preventive treatment with monoclonal antibodies targeting calcitonin gene related piptide (CGRP) or CGRP receptors, or current use of small-molecule CGRP receptor antagonist (e.g. erenumab, fremanezumab, galcaneszumab, atogeptant or rimegepant)
* Changes in treatment with selective serotonin reuptake inhibitors (SSRI) or serotonin norepinephrine reuptake inhibitors (SNRI) within the last two months
* Use of the following medication within 30 days prior to screening:

  * Strong and moderate cytochrome P450 3A4 (CYP3A4) inhibitors, including but not limited to systemic (oral/IV) itraconazole, ketoconazole, fluconazole; erythromycin, clarithromycin, telithromycin; diltiazem, verapamil; aprepitant; cyclosporine; nefazodone; cimetidine; quinine; and HIV protease inhibitors
  * Strong and moderate CYP3A4 inducers, including but not limited to barbiturates (eg, phenobarbital and primidone), systemic (oral/IV) glucocorticoids, nevirapine, efavirenz, pioglitazone, carbamazepine, phenytoin, rifampin, rifabutin, and St. John's wort
  * Inhibitors of the BCRP (breast cancer resistance protein) transporter (eg, rifampicin)
  * Drugs with narrow therapeutic margins (eg, digoxin, warfarin)

Other Exclusions

* Female subjects of childbearing potential with a positive pregnancy test assessed at screening or day 1 by a urine pregnancy test.
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 16 weeks after the last dose of investigational product.
* Female subjects of childbearing potential unwilling to use 1 acceptable method of effective contraception during treatment and for an additional 16 weeks after the last dose of investigational product.
* Evidence of current pregnancy or breastfeeding per subject self-report or medical records
* Subject has known sensitivity to any of the products or components to be administered during dosing.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (e.g, Clinical Outcome Assessments) to the best of the subject and investigator's knowledge.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Pain freedom at 2 hours | 2 hours after initial dose
  Pain freedom will be subjectively rated by the patient in a headache diary

OTHER OUTCOMES:
Absence of the most bothersome symptom (MBS) at 2 hours | 2 hours after initial dose
  Patients are to select their MBS prior to randomization, and then only treat an attack that occurs with the pre-specified MBS. 2 hours after initial dose, patients are to subjectively rate if the MBS have disappeared fully or if it is still present
Relapse | 48 hours after initial dose
  Patients, who were pain free 2 hours after the investigational treatment was administered, are to subjectively evaluate if they experienced reoccurrence of headache of any severity within 48 hours of the intake of given treatment.
Headache intensity | Predose, and 0.5, 1, 1.5, 2, 3, 4, 12, 24 and 48 hours after initial dose
  Headache intensity will be subjectively rated by the patient at predefined timepoints on a 4-point scale where 0 = no headache; 1 = mild headache; 2 = moderate headache; 3 = severe headache.
Rescue medication | 48 hours after initial dose
  The patient will record if they take any rescue medication 2 hours after intake of test medication and within 48 hours
Global evaluation | 48 hours after initial dose
  The patient will subjectively rate their global impression of the test medication based on Likert-type verbal scale (e.g., very poor, poor, no opinion, good, very good)
Associated symptom - nausea | Predose, 2, 4, 8, 12, 24- and 48-hours after initial dose
  The presence or absence of nausea
Associated symptom - photophobia | Predose, 2, 4, 8, 12, 24- and 48-hours after initial dose
  The presence or absence of photophobia
Associated symptom - phonophobia | Predose, 2, 4, 8, 12, 24- and 48-hours after initial dose
  The presence or absence of phonophobia
Adverse events | After the first dose of investigational product and until 48 hours after initial dose.
  Any untowards medical events are to be recorded in the diary by the patients. Furthermore, the patient will be instructed to inform the investigator in such case.

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Prof., Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No